CLINICAL TRIAL: NCT01591408
Title: Placebo-controlled Study of EEG Biofeedback Therapy as an Adjunct Treatment for PTSD, Evaluating Symptoms and EEG Dynamics
Brief Title: EEG Biofeedback Therapy as an Adjunct Treatment for PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: Naval Health Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMCSD.2012.0042
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Results first posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-10

CONDITIONS: PTSD; Anxiety; Trauma; Sleep Disorders
Keywords: EEG biofeedback; neurofeedback; therapy; adjunct
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Wounds and Injuries; Sleep Wake Disorders | interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EEG biofeedback (Experimental): Subjects will receive EEG biofeedback according to their own brain rhythms
  Interventions: Device: EEG biofeedback
- sham EEG biofeedback (Sham Comparator): Subjects will receive feedback according to someone else's brain rhythms collected during a different session.
  Interventions: Device: EEG biofeedback

INTERVENTIONS:
Device: EEG biofeedback — EEG data is collected from the scalp. Data is decomposed in real time and a portion of the signal is fed back to the subject via a vibrating stuffed animal and visual cues.
  Other Names: EEG info device

SUMMARY:
The proposed study, "Placebo-controlled study of EEG biofeedback therapy as an adjunct treatment for PTSD, evaluating symptoms and EEG dynamics", will investigate the brain dynamics associated with PTSD symptom reduction associated with EEG biofeedback therapy or sham EEG biofeedback in addition to treatment as usual at the Naval Medical Center, San Diego (NMCSD) OASIS program.

EEG biofeedback treatment protocols for PTSD and other disorders have been developed and honed by private practice clinicians over the past 25 years, during which EEG biofeedback has become an increasingly popular adjunct therapy.

The reported success of EEG biofeedback as a non-drug intervention with lasting efficacy warrants a clinical study investigating not only symptom reduction, but also the underlying neurobiological mechanism. To this end, we propose a study using high density EEG recordings before and after treatment for PTSD symptoms to determine which brain activities correlate with reported symptom changes.

The proposed study could expand treatment alternatives for servicemen with PTSD. If EEG biofeedback is shown to improve symptom reduction over the placebo controlled condition, it would offer a non-pharmacological intervention that would avoid undesirable side effects, and accelerate recovery compared with the current standard of care.

DETAILED DESCRIPTION:
EEG biofeedback is an emerging alternative approach to treating PTSD, for which there is still insufficient evidence to assume unequivocal clinical utility. However, a 1991 report showed PTSD symptom reduction in 14 subjects receiving EEG biofeedback, as compared to 13 subjects receiving traditional treatment (Peniston, 1991), and a recent case study of 2 PTSD patients receiving EEG biofeedback therapy also showed reduce symptom severity using a newer protocol and device (Othmer, 2009). Another recent study focused on the anxiety symptoms of PTSD and showed that EEG biofeedback significantly reduced anxiety compared to subjects not receiving treatment (Walker, 2009).

EEG biofeedback has also been explored as a treatment for non-PTSD related anxiety disorders, with results showing significant changes in reported anxiety correlated with increased or decreased alpha-frequency (~8-12 Hz) power (Hardt, 1978). Similarly, alpha-frequency EEG biofeedback has been shown to reduce anxiety and to reduce heart rate reactivity to a stressor after 8 sessions of EEG biofeedback training (Rice, 1993). While EEG biofeedback has been shown to significantly change EEG power dynamics (Egner, 2004), it is still unclear if and how EEG biofeedback can effect long-term and complex changes in cognitive and/or emotional functioning.

Some attention has been given to other types of biofeedback for the treatment for PTSD, such as heart rate variability (HRV) biofeedback, which may be relevant in understanding the background of biofeedback with respect to PTSD treatment. While one study reported no difference in symptom reduction between treatment as usual and treatment as usual plus HRV biofeedback (Lande, 2010), a handful of other studies have reported significant associations between HRV changes and PTSD symptoms. Specifically, increased HRV was significantly correlated with PTSD symptom reduction, which was more effective with respiratory sinus arrhythmia (RSA) (which affects HRV) biofeedback than with progressive muscle relaxation (Zucker, 2009). Furthermore, combat-related PTSD subjects showed lower resting HRV than controls, but training with HRV biofeedback increased PTSD subjects' HRV and simultaneously decreased their PTSD symptoms (Tan, 2011). Finally, a quantitative EEG study showed that an acute session of RSA biofeedback was associated with an increase in alpha-band power and reduced higher frequency beta-band power, suggesting a neural impact of RSA training and HRV regulation (Sherlin, 2010).

Summary The proposed study of EEG biofeedback at the OASIS program will not only address the clinical efficacy, but also the brain activations associated with specific symptoms of PTSD through collection of high-density EEG data before and after EEG biofeedback treatment. These data will help elucidate the neural correlates of PTSD symptom expression as well as address the potential efficacy of EEG biofeedback therapy as an adjunct treatment for PTSD-like symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Male,
* active military,
* participating in PTSD program at NMCSD

Exclusion Criteria:

* Seizure disorder.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2012-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Onton, PhD, Principal Investigator — Naval Health Research Center
Locations (1):
- OASIS PTSD program, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EEG Biofeedback | Sham EEG Biofeedback
Started | 36 | 32
Completed | 24 | 24
Not Completed | 12 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EEG Biofeedback | Sham EEG Biofeedback | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (5.2) | 29.4 (5.6) | 29.9 (5.4)
Gender [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 22 | 21 | 43
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Improved Symptom Ratings
Description: Will test whether subjects receiving real EEG biofeedback report decreased anxiety and irritability relative to subjects receiving sham biofeedback. The scale for each rating was a 0-10, with 0 meaning "not at all" and 10 being "extremely" anxious/irritable.
Time Frame: 4 weeks
Population: Subjects were active duty military with PTSD diagnosis currently in residential treatment facility
Measure: Mean (Standard Deviation); unit: Rating on scale
Arm/Group | EEG Biofeedback | Sham EEG Biofeedback
Number analyzed (Participants) | 24 | 24
Rating on scale
  Irritability | -2.62 (2.40) | -1.62 (2.23)
  Anxiety | -2.25 (2.22) | -1.21 (2.23)

ADVERSE EVENTS:
Description: Serious and Other (Not Including Serious) Adverse Events were not collected/assessed
Arm/Group | EEG Biofeedback | Sham EEG Biofeedback
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No